CLINICAL TRIAL: NCT06728514
Title: Comparative Study of Ultrasound Guided Erector Spinae Plane Block vs Ultrasound Guided Paravertebral Block For Post-oprative Analgesia In Patient's After Open Renal Surgeries
Brief Title: Comparative Study of USG Guided ESPB vs USG Guided PVB For Post-op Analgesia In Patient's After Open Renal Surgeries
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sahiwal medical college sahiwal (Other Government)
Collaborators: Department of medical education (Unknown)
Responsible Party: Principal Investigator, Dr. Mujahid jamil, Resident Anaesthesiology, Sahiwal medical college sahiwal
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 98/IRB
Record Dates: First submitted 2024-09-29; First posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Post Operative Analgesia; Hemodynamic (MAP) Stability; Renal Surgeries; Hypertension
Keywords: ESPB; PVB; ASA
MeSH Terms: conditions — Hypertension | interventions — Bupivacaine

STUDY DESIGN:
Intervention Model Description: Group A will receive ESPB and Group B will receive PVB
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GROUP-ESPB (Experimental): Erector spinae plane block
  Interventions: Procedure: Erector spinae plane block group.; Drug: Inj Bupivacaine
- GROUP-PVB (Experimental): Para vertebral block
  Interventions: Procedure: Paravertebral Nerve Block; Drug: Inj Bupivacaine

INTERVENTIONS:
Procedure: Erector spinae plane block group. — In ESPB technique the linear transducer will be placed over the spinous process of the vertebra and a point 3 cm lateral to it are marked at the T10-T11 level before performing the block. Under aseptic precautions, the 23G spinal needle is inserted and advanced perpendicular to the skin in all planes to contact the transverse process of the vertebra. The transverse process of the thoracic vertebra lies at a variable depth of 2-4 cm from the skin depending on the build of the individual. At this point, the needle tip lies between the erector spinae muscle and transverse process. After negative aspiration, local anesthetic is injected in 3-5 ml aliquots. A volume of 20-25 ml of 0.25% bupivacaine will be used for analgesia on each side depending upon the surgery and requirements. The number of attempts will be noted.Time taken to perform block in minutes will be noted from placing transducer to taking out needle after injecting drug in plane.
  Other Names: ESPB
  Arms: GROUP-ESPB
Procedure: Paravertebral Nerve Block — In PVB technique the patient will be placed in the lateral position, and the superior aspect of the T9,T10 and T11 spinous processes will be identified. Under complete aseptic precautions and after skin infiltration with LA, 23G spinal needle will be inserted perpendicular to the skin, with the goal of contacting the tranverse process. Once the TP is contacted, generally at a depth of 2 to 5 cm in adults, the needle is withdrawn into the subcutaneous tissue, redirected in a caudal direction, and then slowly advanced with the purpose of entering the PVS at an approximate depth of 1.0 to 1.5 cm past the initial contact with the TP. After perforating the costotransverse ligament and negative aspiration for blood, air, or spinal fluid,10 mL of 0.25% bupivacaine will be injected at each level superficial to to the pleural line. Displacement of the pleura line anteriorly will be confirmed proper injection of the local anaesthetic solution. The number of attempts will be noted.
  Other Names: PVB
  Arms: GROUP-PVB
Drug: Inj Bupivacaine — Inj Bupivacaine 0.25% (10ml) in both groups
  Other Names: BUPIVACAINE

SUMMARY:
Pain control following open renal surgeries are of utmost importance in order to reduce the chance of chronic pain development, and facilitate early rehabilitation. The erector spinae plane block (ESPB) is a recently developed regional anaesthesia procedure successfully used for different types of surgical procedures including open renal surgeries.

A Comparative cross-sectional study design will be used and patients fulfilling the inclusion criteria will be included that are admitted through the Outpatient department. Patients will be optimized for surgery. A detailed history will be taken regarding the mode of injury, any preexisting disease and previous surgery and finally thorough examination of the patient will be done to rule out any systemic disease. Informed consent will be taken. These patients will be divided into 2 groups by simple lottery method in group A and B.All the data collected will be entered and analyzed by SPSS version 25.0. Age, surgery d.uration, intraoperative heart rate, intraoperative MAP, total postoperative opioid consumption, total intraoperative opiod and isoflurane consumption, time to first required analgesic, and VAS during the first postoperative 24 h will be summarized, according to normality, into mean (± standard deviation [SD]) or median (range). According to data normality, the hypothesis of significant differences between the two studied groups will be challenged using the one-way analysis of variance (with least significant difference correction) or Kruskal-Wallis tests (VAS). Moreover, a p value of < 0.05 will be regarded to be statistically significant

DETAILED DESCRIPTION:
After identifying eligible patients, written consent will be taken from them patients will be counselled about Numeric Rating Scale (NRS) scoring system. A score of 0 will be considered no pain, a score of 1-3 will be considered mild pain, 3-6 will be considered moderate pain and 7-10 as severe pain. Participants will be randomized in a parallel design with a computer-generated assignment to either local anaesthetic ESPB (Group A) or PVB (Group B) in a 1:1 ratio. In pre OP room intravenous access will be obtained and a monitor will be attached and baseline vitals will be measured i.e, blood pressure, heart rate, oxygen saturation, respiratory rate and temperature.Patients will be operated under General anaesthesia monitor will be attached to measure blood pressure, heart rate respiratory rate, oxygen saturation and ECG. Induction will be done with inj. Propofol 2mg/kg, inj. Atracurium 0.5mg/kg; ETT with cuff will be passed and fixed. Inj. Nalbuphine 0.1mg/kg and inj. Paracetamol 10mg/kg will be given for analgesia. Anaesthesia will be maintained by 50:50 mixture of oxygen and nitrous oxide as well as 1-1.5 MAC of Isoflurane and inj. Atracurium 0.1mg/kg boluses on requirement. At the end of the surgical procedures on OT table USG ESPB or PVB will be perfomed.In ESPB technique the linear transducer will be placed over the spinous process of the vertebra and a point 3 cm lateral to it are marked at the T10-T11 level before performing the block. Under aseptic precautions, the 23G spinal needle is inserted and advanced perpendicular to the skin in all planes to contact the transverse process of the vertebra. The transverse process of the thoracic vertebra lies at a variable depth of 2-4 cm from the skin depending on the build of the individual. At this point, the needle tip lies between the erector spinae muscle and transverse process. After negative aspiration, local anesthetic is injected in 3-5 ml aliquots. A volume of 20-25 ml of 0.25% bupivacaine will be used for analgesia on each side depending upon the surgery and requirements. The drug injected in this plane spreads in the longitudinal axis to both cephalad and caudal direction over several levels as the erector spinae fascia extends from nuchal fascia to the sacrum. The number of attempts will be noted. Time taken to perform block in minutes will be noted from placing transducer to taking out needle after injecting drug in plane.In PVB technique the patient will be placed in the lateral position, and the superior aspect of the T9,T10 and T11 spinous processes will be identified. The needle insertion point will be marked approximately 2.5-3 cm lateral from the midline. At these points, Under complete aseptic precautions and after skin infiltration with LA, 23G spinal needle will be inserted perpendicular to the skin, with the goal of contacting the tranverse process. Once the TP is contacted, generally at a depth of 2 to 5 cm in adults, the needle is withdrawn into the subcutaneous tissue, redirected in a caudal direction, and then slowly advanced with the purpose of entering the PVS at an approximate depth of 1.0 to 1.5 cm past the initial contact with the TP. The depth of the PVS has been estimated at 3 to 6 cm from the skin surface. After perforating the costotransverse ligament and negative aspiration for blood, air, or spinal fluid, 10 mL of 0.25% bupivacaine will be injected at each level superficial to the pleural line. Displacement of the pleura line anteriorly will be confirmed proper injection of the local anaesthetic solution. The number of attempts will be noted. Time taken to perform block in minutes will be noted from placing transducer to taking out needle after injecting drug in plane.All the patients will recover from general anaesthesia, inj. Neopyrolate 0.05mg/kg will be given as reversal. Awake extubation will be done. After recovery pain will be assessed at 4, 8, 12 and 24 hours as primary outcome. Postoperative pain will be assessed using NRS ranging from 0 to 10, on which 0 means no pain and 10 will show worst pain. A higher score will indicate the worst outcome. A score of 0 will be taken as no pain, a score of 1-3 will be considered mild pain, 3-6 will be considered moderate pain, and 7-10 as severe pain. The nurse will assess the outcome, and both the nurse and patients will be blind and unaware about the group they will in to prevent any bias in the study. Secondary outcomes will include, ease of performance, rescue analgesia time and opiod sparing effect.

For pain-relief medications, inj. Tramadol 1mg/kg will be given to the patient when NRS score is 4 or more. For bradycardia inj. Atropine 0.01mg/kg will be given. For nausea complain, ondansetron will be administered with the first dose of 4 mg followed by 1 mg if required. No prophylactic antiemetics will be administered.

ELIGIBILITY:
Inclusion Criteria:

Both Genders Age between 18 years to 60 years. BMI ≤ 30 kg/m2 ASA I or ASA II

Exclusion Criteria:

Patients who do not give consent. Relevant drug allergy. Pregnancy Alcohol or drug abuse. Infection at the site of injection. Taking of pain medications within 24 h before surgery. Chronic hepatic or renal failure. Deranged coagulation profile

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2024-01-11 (Actual); Primary Completion 2024-07-09 (Actual); Study Completion 2024-08-09 (Actual)

PRIMARY OUTCOMES:
Post Op Analgesia | From performance of block to first rescue analgesia in 24 hours post operatively.
  Duration of post op analgesia.

CONTACTS AND LOCATIONS:
Overall Officials: Adeel Riaz, MD, Study Director — Sahiwal Teaching Hospital, Sahiwal
Locations (1):
- Sahiwal Medical College,Sahiwal, Sahiwal, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Data will be available on request
Supporting Information: Study Protocol, SAP, ICF
Time Frame: August 2024
Access Criteria: On Demand